CLINICAL TRIAL: NCT04891666
Title: A Clinical Trial to Evaluate the Efficacy and Safety of Lactobacillus Plantarum DSM 33464 (SmartGuard®) on Blood Lead Levels in Children
Brief Title: A Trial to Evaluate the Efficacy and Safety of Lactobacillus Plantarum DSM 33464 on Blood Lead Levels in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novozymes A/S (Industry)
Collaborators: Beijing Children's Hospital (Other); Baoding Children's Hospital (Other); Xuzhou Children Hospital (Other); Chengdu Women's and Children's Central Hospital (Other); Children's Hospital of Heibei Province (Unknown); Beijing Clinical Service Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NZ-GHSG-2020-02
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Elevated Blood Lead Levels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus plantarum DSM 33464 (Experimental): 1 sachet of Lactobacillus plantarum DSM 33464 (2 g) and 1 sachet of supplement YingKangWei per day for 12 weeks
  Interventions: Dietary Supplement: Lactobacillus plantarum DSM 33464
- placebo (Placebo Comparator): 1 sachet of placebo (2 g) and 1 sachet of supplement YingKangWei per day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum DSM 33464 — 1 sachet SmartGuard® per day for 12 weeks
  Other Names: SmartGuard®
  Arms: Lactobacillus plantarum DSM 33464
Dietary Supplement: Placebo — 1 sachet of placebo per day for 12 weeks
  Arms: placebo

SUMMARY:
The study is a parallel, randomized, double-blind, placebo controlled clinical trial will evaluate the effect of Lactobacillus plantarum DSM 33464 on reduction of Blood lead levels and general well-being of children.

ELIGIBILITY:
Inclusion Criteria:

The subjects who meet all of the following selection criteria can participate in this study:

1. Children age 3-12 years
2. BLL 35-249 µg/L
3. Subjects, their parents or legal guardians are able and willing to comply with research guidance
4. Subject's parents or legal guardians sign written informed consent.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria may not participate in this study:

1. Diagnosed with nervous system diseases, genetic and metabolic diseases, endocrine diseases, lung diseases, severe or unstable cardiovascular diseases, clinically significant kidney or liver diseases, blood system diseases, any other clinically significant diseases and Other investigators judge that the participation of subjects in the study will increase the risk of the subjects' diseases;
2. History of infection or organ transplantation of human immunodeficiency virus or other acquired congenital immunodeficiency diseases;
3. Take probiotic products in the last two weeks
4. Known or suspected sensitivity or allergy to food or any constituents tested in the trial
5. Participation in another clinical trial or food study 4 weeks prior and during the trial

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Reduction of blood lead levels | 12 weeks
  Difference in reduction of blood lead level between the experimental group and the placebo group at week 12 compared with baseline

SECONDARY OUTCOMES:
Reduction of blood lead levels | 4 and 8 weeks
  Compared with the baseline, the difference between the reduction of the blood lead level in the experimental group and the placebo group at the 4th and 8th week
Reduction of urine lead levels | 4, 8 and 12 weeks
  Compared with baseline, the difference between the reduction of urine lead levels in the experimental group and the placebo group at the 4th, 8th, and 12th week
Improvement of common trace elements-Ca,Zn,Cu,Mg,Fe in the blood | 4, 8 and 12 weeks
  Compared with baseline, the difference between the improvement of common trace elements Ca,Zn,Cu,Mg,Fe in the blood of the experimental group and the placebo group at the 4th, 12th and 24th week

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Baoding children's hospital, Baoding, Hebei
  - Children's Hospital of Heibei Province, Shijiazhuang, Hebei
  - Xuzhou children's Hospital, Xuzhou, Jiangsu
  - Chengdu women's and children's Central Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji W, Saulnier DM, Zhang L, Liu J, Gao J, Wang X, Holz C, Liang A, Tan HT. Effects of Lactiplantibacillus plantarum DSM 33464 in children with elevated blood lead levels: a randomized, double-blind, placebo-controlled study. Front Nutr. 2025 Sep 1;12:1641839. doi: 10.3389/fnut.2025.1641839. eCollection 2025. PMID 40959702